CLINICAL TRIAL: NCT01041547
Title: Vitamin D, Vascular Function, and Insulin Sensitivity in Adults [The VIVID Study
Brief Title: Vascular Function, Insulin Sensitivity, and Vitamin D
Acronym: VIVID
Status: Completed | Type: Observational
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Ambika Ashraf, M.D., Associate Professor, University of Alabama at Birmingham
Other Study IDs: F091023002
Record Dates: First submitted 2009-12-28; First posted 2009-12-31 (Estimated); Last update posted 2014-01-14 (Estimated); Status verified 2014-01

CONDITIONS: Insulin Sensitivity; Flow-mediated Dilation; Arterial Stiffness
Keywords: Insulin sensitivity; Vascular function; Flow-mediated dilation; Arterial stiffness; Glucose tolerance; Hypertension
MeSH Terms: conditions — Insulin Resistance; Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Seum
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Healthy adults: healthy adults with BMI below 32, between ages 19-60 yrs, both males and females

SUMMARY:
The overall objectives of this study are to examine the relationships between circulating vitamin D, insulin sensitivity, and multiple indices of vascular function and to examine whether vitamin D deficiency in African Americans (AA) and White Hispanics (WH) is responsible for ethnic differences in insulin sensitivity and hypertension in AA, WH and European Americans (EA), as well as mechanisms underlying the association between insulin resistance and blood pressure. We hypothesize that 1) serum 25(OH)D is associated with insulin sensitivity and vascular functioning, independent of adiposity, 2) lower insulin sensitivity and vascular functioning in AA and WH relative to EA is due to lower circulating 25(OH)D in AA, and 3) the relationship between insulin resistance and vascular dysfunction is mediated by 25(OH)D.

Acronyms: African American (AA), European American (EA), White Hispanics (WH), Serum 25-hydroxy vitamin D (25()H)D, Body mass index (BMI), Alabama (AL).

ELIGIBILITY:
Inclusion Criteria:

* African American (AA), White Hispanic (WH), and European American (EA) race
* Ages 19-60 years
* Negative urine pregnancy test
* No evidence of diabetes
* Not on medications that can affect vascular functioning or insulin sensitivity

Exclusion Criteria:

* BMI > 32 kg/m2
* Diabetes or any chronic diseases
* Use of medication(s) known to influence body composition, vascular function, or glucose metabolism
* Regular smoking
* Regular use of illegal drugs and pregnancy

Ages: 19 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: * Healthy adults with BMI below 32
  * Both males and females
  * Ages 19-60 years
  * Race: African Americans, White Hispanics, European Americans
Sampling Method: Non-Probability Sample
Enrollment: 63 (Actual)
Dates: Start 2009-12; Primary Completion 2012-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Insulin sensitivity | Cross sectional study: at first study visit

SECONDARY OUTCOMES:
Vascular function | Cross sectional study: at second study visit, within 2 weeks of first study visit

CONTACTS AND LOCATIONS:
Overall Officials: Ambika Ashraf, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama, Birmingham, Alabama, United States

REFERENCES:
- [Derived] Alvarez JA, Gower BA, Calhoun DA, Judd SE, Dong Y, Dudenbostel T, Scholl J, Ashraf AP. Serum 25-hydroxyvitamin D and Ethnic Differences in Arterial Stiffness and Endothelial Function. J Clin Med Res. 2012 Jun;4(3):197-205. doi: 10.4021/jocmr965w. Epub 2012 May 15. PMID 22719806